CLINICAL TRIAL: NCT02593071
Title: A Phase II Randomized, Observer-Blind, Placebo-Controlled Study to Evaluate the Immunogenicity and Safety of a Respiratory Syncytial Virus (RSV) Recombinant F Nanoparticle Vaccine in Healthy Older Adult Subjects Previously Treated With the Same Vaccine, or Placebo, in the Prior Year; and to Estimate the Incidence Rate of RSV Disease and Vaccine Efficacy in Subjects Based on Their RSV F Vaccine Experience Over Two Consecutive Years.
Brief Title: Safety and Immunogenicity of the RSV-F Vaccine in Older Adults Previously Treated With the Same Vaccine or Placebo in the Prior Year.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RSV-E-202
Record Dates: First submitted 2015-10-22; First posted 2015-10-30 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Syncytial Virus (RSV)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group A (Experimental): RSV-F Vaccine ( 0.5mL Injection)
  Interventions: Biological: RSV-F Vaccine
- Treatment Group B (Placebo Comparator): Phosphate Buffer Placebo (0.5mL Injection)
  Interventions: Biological: Phosphate Buffer Placebo

INTERVENTIONS:
Biological: RSV-F Vaccine
  Arms: Treatment Group A
Biological: Phosphate Buffer Placebo
  Arms: Treatment Group B

SUMMARY:
This study will enroll subjects who received the RSV F vaccine or placebo in the earlier study (RSV-E-201, Year 1) and re-randomize them to receive either vaccine or placebo in a second season. This design will permit evaluation of the safety and immunogenicity of revaccination in a second RSV season, and the safety and immunogenicity of revaccination over two years.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥60 years of age who are veterans of the RSV-E-201 clinical trial and who are ambulatory and live in the community or in residential facilities which provide minimal assistance, such that the subject is primarily responsible for self-care and activities of daily living. Subjects may have one or more chronic medical diagnoses, but should be clinically stable as assessed by:

   * Absence of changes in medical therapy within one month due to treatment failure or toxicity,
   * Absence of medical events qualifying as SAEs within two months, and
   * Absence of known, current, life-limiting diagnoses that, in the opinion of the investigator, render survival to trial completion unlikely.
2. Willing and able (on both a physical and cognitive basis) to give informed consent prior to study enrollment.
3. Able to comply with study requirements, including access to transportation for study visits. The investigator may use his/her discretion to assess potential ability and willingness to comply based on performance in the prior trial, RSV-E-201.
4. Access to inbound and outbound communication by telephone with caregivers and study staff.

Exclusion Criteria:

1. Participation in research involving investigational product (drug / biologic / device) within 45 days before planned date of first vaccination, with the exception of participation in the preceding study RSV-E-201.
2. History of a serious reaction to any prior vaccination, or Guillain-Barré syndrome (GBS) within 6 weeks of any prior influenza immunization, or withdrawal from the preceding RSV-E-201 clinical trial due to an adverse event deemed test article-related or at the advice of the investigator.
3. Receipt of any vaccine other than IIV in the 4 weeks preceding the study vaccination; or any RSV vaccine at any time unless administered in the preceding study, RSV-E-201.
4. Any known or suspected immunosuppressive condition, acquired or congenital, as determined by history and/or physical examination.
5. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted.
6. Administration of immunoglobulins and/or any blood products within the 3 months preceding the administration of the study vaccine or during the study.
7. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever, or an oral temperature ≥38.0°C on the planned day of vaccine administration).
8. Known disturbance of coagulation. Potential subjects receiving aspirin, clopidogrel, prasugrel, dipyridamole, dabigatran, apixaban, rivaroxaban or warfarin under good control for cardiovascular prophylaxis or prophylaxis of thromboembolic disease or stroke in the setting of atrial fibrillation will NOT be excluded.
9. Suspicion or recent history (within one year of planned vaccination) of alcohol or other substance abuse.
10. Any condition that in the opinion of the investigator would pose a health risk to the subject if enrolled or could interfere with evaluation of the vaccine or interpretation of study results (including neurologic, cognitive, or psychiatric conditions deemed likely to impair the quality of study compliance or safety reporting).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1330 (Actual)
Dates: Start 2015-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Serum IgG antibody concentrations as ELISA units (EUs) specific for the F protein antigen. | Day 0 to Day 364
  Derived/calculated endpoints based on these data will include:
  * Geometric mean concentration as EU (GMEU)
  * Geometric mean ratio (GMR)
  * Seroresponse rate (SRR)
  * Proportion of subjects with two (2)- and 4-fold seroconversion rates ( SCR2 and SCR4, respectively)
Numbers and percentages of subjects with solicited local and systemic AEs | Day 0 to Day 364
  Solicited local and systemic AEs over the seven days post-injection; and all adverse events, solicited and unsolicited, over 56 days post-dosing (Year 2). In addition, MAEs, SAEs, and SNMCs will be collected for 1 year (approximately 364 days) post-dosing

SECONDARY OUTCOMES:
Palivizumab-competitive antibody (PCA) expressed as µg/mL as detected in a competitive ELISA | Day 0 to Day 182
  Summarized by:
  * Geometric mean concentrations (GMC)
  * Geometric mean ratio (GMR)
  * Proportion of subjects with two (2)- and 4-fold seroconversion rates ( SCR2 and SCR4, respectively)
Neutralizing antibody titer to at least one RSV/A and one RSV/B strain. | Day 0 to Day 182
  Summarized by:
  * Geometric mean titer (GMT)
  * Geometric mean ratio (GMR)
  * Proportion of subjects with two (2)- and 4-fold seroconversion rates ( SCR2 and SCR4, respectively)

OTHER OUTCOMES:
Number and percentages of subjects fulfilling the definitions of RSV-associated respiratory disease and/or RSV-lower respiratory tract disease in various treatment groups. | Day 0 to Day 182
Number and percentages of subjects with respiratory illnesses for which a non-RSV viral respiratory pathogen (with or without concurrent RSV infection) is identified by RT-PCR. | Day 0 to Day 182

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (10):
- United States (10):
  - Nothern California Clinical Research, Redding, California
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Rapid Medical Research, Cleveland, Ohio
  - Clinical Research Associates, Nashville, Tennessee
  - Research Across America, Dallas, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Group Health Research Institute, Seattle, Washington
  - Marshfield Clinical Research Foundation, Wausau, Wisconsin